CLINICAL TRIAL: NCT05974332
Title: Serum Oncostatin M in Ulcerative Colitis Patients and Its Relation to Severity and Acute Exacerbation
Brief Title: Oncostatin M in Ulcerative Colitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, mohamed gamal mohamed abdel aleem, Doctor, Beni-Suef University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Beni-Suefu
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulcerative colitis Patients (Active Comparator): 45 Patients with UC. The diagnosis of UC will be based on endoscopic finding and histopathological finding
  Interventions: Diagnostic Test: Oncostatin M
- Control (Active Comparator): 45 apparently healthy subjects as controls who were not UC
  Interventions: Diagnostic Test: Oncostatin M

INTERVENTIONS:
Diagnostic Test: Oncostatin M — Test to diagnosis of Ulcerative colitis

SUMMARY:
Ulcerative colitis (UC) is a refractory disease characterized by symptoms such as diarrhea, bloody stools, and abdominal pain with repeated relapses and remissions.

DETAILED DESCRIPTION:
Evaluation of UC activity is important, and endoscopic evaluations of mucosal inflammation can facilitate subsequent prognostication. On the basis of these considerations, achievement of mucosal healing is important in inflammatory bowel disease (IBD), and evaluation of IBD using endoscopy is extremely important. However, endoscopic examinations are associated with problems such as physical burden to the patient, cost, and risk of complications.

Thus, to avoid the need for frequent endoscopy, noninvasive biomarkers that accurately reflect the endoscopic activity of UC have emerged, and fecal calprotectin (FC) and the fecal immunochemical occult blood test (FIT) are being widely used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years and <80 years, of both gender who diagnosed to have UC and given the consent for participation in the study

Exclusion Criteria:

* 1- Any patient with systemic inflammation as Bronchial asthma. 2- History of cancer or tumor. 3- Autoimmune disease such as rheumatoid arthritis and systemic lupus erythematous

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Identify if oncostatin M is a good marker | 6 months
  Diagnosis of Ulcerative colitis and follow up